CLINICAL TRIAL: NCT00204997
Title: Preservation of Ovarian Function Via Laparoscopic Transposition in Patients With Locally Advanced Squamous Cell Carcinoma of the Cervix
Brief Title: Preservation of Ovarian Function Via LOT in Squamous Cell Carcinoma of the Cervix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO02702; 2002-255; A532820 (Other: UW Madison); SMPH/OBSTET & GYNECOL/OBSTET (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2008-06

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Squamous Cell; Laparoscopy; Ovarian Function
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Laparoscopic Ovarian Transposition
  Interventions: Procedure: Laparoscopic ovarian transposition

INTERVENTIONS:
Procedure: Laparoscopic ovarian transposition — Laparoscopic ovarian transposition

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and efficacy of laparoscopic ovarian transposition in women less than 40 years of age with locally advanced cervical squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Stages iB-iiiB squamous cell carcinoma of the cervix

Exclusion Criteria:

* Evidence of ovarian involvement on MRI
* Evidence of uterine involvement on MRI
* Evidence of distant mets on MRI

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2002-09; Primary Completion 2005-09 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Menopause | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David M Kushner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/